CLINICAL TRIAL: NCT00562042
Title: Risk Stratification for Patients Presenting With Acute Pulmonary Embolism (PE)
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to slow accrual of patients.
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 04-10006
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; risk stratification; prognosis; troponin; Brain natriuretic peptide; echocardiogram
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with acute pulmonary embolism were enrolled in this study.

SUMMARY:
Hypothesis: Increases in CRP, trop T, and BNP values will correlate significantly with right heart failure on echocardiogram and with mortality, ICU stay, hospital stay, and escalations in care.

1. Evaluate whether CRP, trop T, and BNP correlate significantly with right heart failure on echocardiogram.
2. Evaluate whether CRP, trop T, BNP, and echocardiogram correlate significantly with clinical outcomes: mortality, ICU stay, hospital stay, and escalations in care.
3. Compare each test's correlation with clinical outcomes to the others, to determine which test provides the best risk ratio.
4. Compare each trop T value's correlation with echo findings and clinical outcomes to determine the optimal time to draw trop T levels on a patient presenting with acute PE.
5. These tests will not be used in an attempt to establish a diagnosis of PE.

DETAILED DESCRIPTION:
Purpose: This study will help us to determine whether laboratory tests used to evaluate cardiac function and blood flow (troponin T (trop T), C-reactive protein (CRP), and brain-natriuretic peptide (BNP)) correlate with findings on echocardiogram and with meaningful clinical outcomes when patients present with acute pulmonary embolism (PE). We will be studying these tests for prognostic purposes only, in patients with an established diagnosis of PE.

Research design: Prospective cohort study Methodology: Patients diagnosed with acute PE (see exclusion and inclusion criteria below) will be offered enrollment in the study. Once enrolled, he/she will then have a trans-thoracic echocardiogram (TTE) performed by a member of the cardiology service who will not be aware of the patient's clinical status, co-morbidities, or lab results (other than knowing that the patient has been diagnosed with acute PE). The patient will then have trop T, CRP, and BNP levels drawn (or added to laboratory tests that have already been drawn), which will be ordered by a member of the research team. CRP and BNP will be drawn only once, while trop T levels will be drawn every 4 hours for the first 24 hours, and every 8 hours from 24 to 48 hours. The primary team managing the patients will be privy to both the additional laboratory values ordered by the research team and the results of the TTE.

Each patient will be followed for the remainder of their hospital stay by a member of the research team. The following outcomes will be recorded: deaths, length of ICU stay, length of hospital stay, and escalations in care (pressor support, cardiopulmonary resuscitation (CPR), administration of thrombolytics, mechanical ventilation, ICU transfer).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Acute PE (diagnosed by pulmonary angiogram, Computed tomography using the DVT/PE protocol, Ventilation/Perfusion (V/Q) scan read as high probability by the radiologist, or (+) lower extremity Doppler ultrasound with symptoms consistent with PE)

Exclusion Criteria:

* Hemodynamic instability (BP < 90/60, IV pressor support) on admission
* Acute respiratory failure on admission
* Treatment with thrombolytic therapy prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2004-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
mortality | In hospital mortality.

SECONDARY OUTCOMES:
Escalations in care - thrombolysis, CPR, mechanical intubation, transfer to ICU, IV vasopressor administration | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Holley, MD, Principal Investigator — Walter Reed Army Medical Center